CLINICAL TRIAL: NCT03542253
Title: Combined Diagnosis of CT and Exosome in Early Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, gongjianping, Combined diagnosis of CT and exosome in early lung cancer, Second Affiliated Hospital of Soochow University
Other Study IDs: 123456
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Early Lung Cancer
Keywords: Early lung cancer,ground-glass nodule,CT,exosome
MeSH Terms: conditions — Lung Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (17):
- Age
- Sex
- triglyceride
- Lipoprotein
- CT: Target Reconstruction
- micorRNA-A Plasma exocrine
- micorRNA-A Paracancerous tiusse
- pathologic diagnosis
  Interventions: Procedure: Surgery
- hemolysis
- ct-DNA
- micorRNA-A in plasma
- Sample quality control
- positive
- negative
- micorRNA-R in plasma
- micorRNA-R in Plasma exocrine
- Surgery

INTERVENTIONS:
Procedure: Surgery — After surgical treatment, pathological specimens were extracted to obtain pathological results
  Groups: pathologic diagnosis

SUMMARY:
This experiment has now collected 50 cases, all through CT chest scans and blood exosome detection. Twenty-two patients underwent surgical treatment and 14 tissue specimens were examined for cancer and paracancerous tissue exosomesWe found that exosomal micor-A was highly expressed in early stage lung cancer tissues and was significantly higher than paracancerous tissues. The micor-A in the adjacent tissues was significantly higher than that in peripheral blood exosomes

ELIGIBILITY:
Inclusion Criteria:1. At least 18 years of age, male or female; 2. No patients with acute disease; 3. Chest or LDCT examination for the first time found 5-30mm pulmonary nodule patients, and ruled out disseminated tuberculosis; 4. Past pulmonary nodes Festival failed to diagnose. 5. Have not received a history of surgical treatment of the lungs; 6. Patients who have not received targeted drugs, biological treatments, immunosuppressive agents, and modulators; 7. No organ transplants; 8. Signed informed consent before undergoing clinical studies Consent and adherence to the research protocol.

-

Exclusion Criteria:1. Pulmonary nodules have been treated surgically (considering that surgery has been performed to interfere with the study); 2. History of organ transplants such as lung transplantation (consider the use of allogeneic genes and immunosuppressive agents); 3. Pregnancy or lactation (consider Failure to perform regular CT follow-up and fetal component effects. 4. Known HIV-positive or only AIDS-related diseases (taking into account interference with the use of immune drugs); 5. Being targeted drugs, immunosuppressive agents, immunomodulators, biotherapies Patients; 6. Active pulmonary tuberculosis (consider infectious and referral missing factors); 7. RNA-like viral infections: such as SARS, HIV, hepatitis virus (except for hepatitis B, the other four are all RNA viruses), influenza virus, Bird flu virus, H5N1, Ebola, measles, etc. 8. Various blood system diseases such as leukemia, lymphoma, aplastic anemia, myelodysplastic syndrome, anemia, hemolysis, hemophilia, DIC, etc. 9. Recent history of blood transfusion (within 3~6 years) and potential for blood transfusion; 10. Patients with neurological disorders and mental disorders unable to cooperate; 11. Emergency treatment for acute and severe diseases; 12. No Willing to sign a written informed consent and follow the study protocol before they are willing to conduct clinical research; 13. The presence of the patient may interfere with any psychological, family, social or geography conditions that obey the requirements of the research protocol or the follow-up procedure. Discuss these conditions with the patient before entering the study.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: From November 2017 to June 2019, there were nodules on the lungs, both men and women, and patients of the same age who had CT target reconstruction and miRNA and ctDNA detection at the same time had complete follow-up data.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-05-20 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
exosome in cancer tissue and para cancerous tissue | one year
  exosomal micor-A was highly expressed in early stage lung cancer tissues